CLINICAL TRIAL: NCT00383383
Title: To Compare the Immunogenicity & Safety of GSK Biologicals New Adjuvanted Hepatitis B Vaccine to a Double Dose of Engerix™-B, in Pre-Haemodialysis/Haemodialysis Patients (≥15 Years of Age)
Brief Title: Comparison of Adjuvanted Hepatitis B Vaccine to Double Dose of Engerix™-B in Pre- /Haemodialysis Patients Aged ≥15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/042
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B

INTERVENTIONS:
Biological: Hepatitis B adjuvanted vaccine
Biological: Engerix-B

SUMMARY:
Comparison of adjuvanted hepatitis B vaccine to double dose of Engerix™-B in pre- /haemodialysis patients aged ≥15 years.

ELIGIBILITY:
Inclusion Criteria:

* A male or female > = 15 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/ from the parents or guardians of the subject.
* Seronegative for anti-HBs antibodies, anti-HBc antibodies & Hepatitis B Surface antigen (HBsAg).
* If the subject was a female, she was of non-childbearing potential or, if of childbearing potential, she had to be abstinent or use adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination.
* Pre-haemodialysis patient* or a patient on haemodialysis.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine during the study period or within 30 days preceding the first dose of study vaccine.
* Previous vaccination against hepatitis B.
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within 6 weeks. Pregnant or lactating female
* Clinically abnormal ALT/AST values (> 3 times normal values)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141
Dates: Start 1999-12

PRIMARY OUTCOMES:
Anti-HBs seroprotection rates at Month 12.

SECONDARY OUTCOMES:
Solicited symptoms, unsolicited symptoms and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Clinical Trials Call Center, Hradec, Králové, Czechia
- GSK Clinical Trials Call Center, Kuala Lumpur, Malaysia
- GSK Clinical Trials Call Center, Málaga, Spain